CLINICAL TRIAL: NCT01542034
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study of ATX-101 (Sodium Deoxycholate Injection) Versus Placebo for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Phase 3 Study of Deoxycholic Acid Injection (ATX-101) Versus Placebo for the Reduction of Localized Subcutaneous Fat in the Submental Area
Acronym: REFINE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATX-101-11-22
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deoxycholic Acid Injection (Experimental): Participants received deoxycholic acid 2 mg/cm² administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Deoxycholic acid injection
- Placebo (Placebo Comparator): Participants received placebo administered in 0.2 mL injections, up to 10 mL per treatment session at intervals of approximately 1 month for up to a maximum of 6 treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deoxycholic acid injection — Formulated as an injectable solution containing deoxycholic acid at a concentration of 10 mg/mL.
  Other Names: ATX-101; Kybella
  Arms: Deoxycholic Acid Injection
Drug: Placebo — Phosphate buffered saline placebo for injection
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of deoxycholic acid injection in the reduction of submental fat (fat below the chin).

ELIGIBILITY:
Inclusion Criteria:

1. Submental fat graded by the investigator as 2 or 3 using the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and graded by the subject as 2 or 3 using the Patient-Reported Submental Fat Rating Scale (PR-SMFRS) as determined on Visit 1 (within 28 days before randomization).
2. Dissatisfaction with the submental area expressed by the subject as a rating of 0, 1, or 2 using the Subject Self Rating Scale (SSRS) as determined on Visit 1 (within 28 days before randomization).
3. Males and nonpregnant, nonlactating females 18 to 65 years of age, inclusive, on the day of randomization (Visit 2). Females of childbearing potential must have a negative human chorionic gonadotropin (hCG) test result within 28 days before Visit 2 and agree to practice adequate contraception, in the judgment of the investigator, during the course of the study. Females of childbearing potential who are not sexually active need not practice contraception.
4. History of stable body weight, in the judgment of the investigator, for at least 6 months before randomization.
5. Expected to understand and agree to comply with the visit schedule and all protocol-specified tests and procedures and agreement by the subject to refrain from making significant changes, in the judgment of the investigator, to his or her dietary or exercise habits during the course of the subject's participation.
6. Agreement to forego any treatment or behavior (e.g., unshaven facial hair) during the subject's participation in the study that may affect the assessments of the submental area.
7. Medically able to undergo the administration of study material determined by clinical and laboratory tests obtained within 28 days before randomization for which the investigator identified no clinically significant abnormality.
8. Signed informed consent obtained before any study-specific procedure is performed.

Exclusion Criteria:

1. History of any intervention to treat submental fat (e.g., liposuction, surgery, or lipolytic agents).
2. History of trauma associated with the chin or neck areas that in the judgment of the investigator may affect evaluation of safety or efficacy of treatment.
3. A Submental Skin Laxity Grade (SMSLG) of 4 or other anatomical feature (e.g., predominant subplatysmal fat, loose skin in the neck or chin area, prominent platysmal bands), as assessed within 28 days before randomization, for which reduction in submental fat may, in the judgment of the investigator, result in an aesthetically unacceptable outcome.
4. Evidence of any cause of enlargement in the submental area (e.g., thyroid enlargement, cervical adenopathy) other than localized submental fat.
5. Body mass index of > 40.0 as determined on Visit 1.
6. History or current symptoms of dysphagia.
7. A result on coagulation tests (PT, PTT) obtained within 28 days before randomization that indicates the presence of any clinically significant bleeding disorder.
8. Any medical condition (e.g., respiratory, cardiovascular, hepatic, neurological disease, or thyroid dysfunction) that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or give informed consent.
9. Treatment with radio frequency, laser procedures, chemical peels, or dermal fillers in the neck or chin area within 12 months before randomization.
10. Treatment with botulinum toxin injections in the neck or chin area within 6 months before randomization.
11. History of sensitivity to any components of the study material
12. History of sensitivity to topical or local anesthetics (e.g., lidocaine, benzocaine, procaine).
13. Previous randomization in this study or previous participation in a Kythera-sponsored ATX 101 trial.
14. Treatment with an investigational device or agent within 30 days before randomization.
15. For centers selected to conduct magnetic resonance imaging (MRI) evaluations, any subject with the presence of any condition that would render a subject unsuitable for MRI evaluation (e.g., claustrophobia), or metals in the body that would interfere with MRI acquisition (e.g., nonremovable metal appliances in the mouth such as silver or gold caps, pacemakers, metal joints).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, MD, PhD, Study Director — Kythera Biopharmaceuticals, Inc
Locations (31):
- United States (27):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Beverly Hills, California
  - Investigational Site, Irvine, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Oceanside, California
  - Investigational Site, San Diego, California
  - Investigational Site, New Haven, Connecticut
  - Investigational Site, Washington D.C., District of Columbia
  - Investigational Site, Miami Beach, Florida
  - Investigational Site, West Palm Beach, Florida
  - Investigational Site, Atlanta, Georgia
  - Investigational Site, Snellville, Georgia
  - Investigational Site, Arlington, Illinois
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Evansville, Indiana
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Glenn Dale, Maryland
  - Investigational Site, Hunt Valley, Maryland
  - Investigational Site, Rockville, Maryland
  - Investigational Site, West Bloomfield, Michigan
  - Investigational Site, Fridley, Minnesota
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, New York, New York
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Charlottesville, Virginia
  - Investigational Site, Spokane, Washington
- Canada (4):
  - Investigational Site, Peterborough, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Montreal, Quebec
  - Investigational Site, Vancouver, B.C.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at 35 investigational centers in the United States (US) and Canada.
Period: Overall Study
Arm/Group | Deoxycholic Acid Injection | Placebo
Started | 256 | 250
Received Treatment | 256 | 249
Completed | 226 (Participants who completed long-term follow-up 24 weeks after the last treatment) | 227 (Participants who completed long-term follow-up 24 weeks after the last treatment)
Not Completed | 30 | 23
Not completed — Consent Withdrawn (Subject Convenience) | 20 | 12
Not completed — Administrative decision | 0 | 3
Not completed — Subject Noncompliance | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Deoxycholic Acid Injection | Placebo | Total
Number analyzed (Participants) | 256 | 250 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (9.30) | 49.4 (9.33) | 49.5 (9.30)
Age, Customized [Number; unit: participants]
  18 - 50 years | 122 | 121 | 243
  51 - 65 years | 134 | 129 | 263
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 208 | 421
  Male | 43 | 42 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  White | 218 | 227 | 445
  Black or African American | 24 | 13 | 37
  Asian | 7 | 5 | 12
  American Indian or Alaskan Native | 0 | 2 | 2
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Multiple | 2 | 0 | 2
  Other | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 28 | 17 | 45
  Non-Hispanic or Latino | 228 | 233 | 461
Weight [Mean (Standard Deviation); unit: kg] — Data available for 256 and 249 participants in each treatment group respectively
  kg | 81.15 (14.549) | 80.98 (14.296) | 81.07 (14.411)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Data available for 256 and 249 participants in each treatment group respectively
  kg/m² | 29.23 (4.406) | 29.26 (4.281) | 29.25 (4.340)
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type is a numerical classification schema for human skin color and typical response to ultraviolet (UV) light:
  * Type I: Pale white skin, blue/hazel eyes, blond/red hair; Always burns, does not tan.
  * Type II: Fair skin, blue eyes; Burns easily, tans poorly.
  * Type III: Darker white skin; Tans after initial burn.
  * Type IV: Light brown skin; Burns minimally, tans easily.
  * Type V: Brown skin; Rarely burns, tans darkly easily.
  * Type VI: Dark brown or black skin; Never burns, always tans darkly.
  participants
    I - III | 180 | 187 | 367
    IV - VI | 76 | 63 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Composite 1-grade Response
Description: A composite 1-grade response is defined as at least a 1-grade improvement from Baseline on both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) 12 weeks after the last treatment.
  The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
  The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0-4) with 0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Intent-to-treat (ITT) population; missing values were imputed using a multiple imputation process.
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection | Placebo
Number analyzed (Participants) | 256 | 250
percentage of participants | 70.0 | 18.6
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection vs Placebo; The primary analysis was satisfied if both null hypotheses (there is no treatment difference in 1-grade or 2-grade response rate) were rejected in favor of the two-tailed alternative at the 0.05 level of significance for both primary efficacy endpoints, and the response rates were higher for the deoxycholic acid injection treatment group than the placebo group. Because both hypotheses must be rejected, the type I error was preserved when testing the primary endpoints; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) method stratified by pooled study center; Risk Ratio (RR) = 3.702, 95% CI 2-sided [2.808 to 4.880] — A risk ratio greater than 1 favors deoxycholic acid injection treatment, and between 0 and 1 favors placebo

2. Primary Outcome: Percentage of Participants Who Achieved a Composite 2-grade Response
Description: A composite 2-grade response is defined as at least a 2-grade improvement from Baseline on both the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS) and Patient-Reported Submental Fat Rating Scale (PR-SMFRS) 12 weeks after the last treatment.
  The CR-SMFRS score is based on the investigator's clinical evaluation of the participant, where submental fullness is scored on a 5-point ordinal scale (0-4) with 0 = absent, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
  The PR-SMFRS is based on the participant's response to the question "How much fat do you have under your chin right now?" answered on a 5-point ordinal scale (0-4) with 0 = no chin fat at all, 1 = a slight amount of chin fat, 2 = a moderate amount of chin fat, 3 = a large amount of chin fat, and 4 = a very large amount of chin fat.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Intent-to-treat population; missing values were imputed using a multiple imputation process.
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection | Placebo
Number analyzed (Participants) | 256 | 250
percentage of participants | 13.4 | 0.0
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH method stratified by pooled study center

3. Secondary Outcome: Percentage of Participants With a Magnetic Resonance Imaging (MRI) Response
Description: An MRI responder is a participant who exhibited at least a 10% reduction in submental fat volume as measured by MRI from Baseline to 12 weeks after last treatment. Magnetic resonance imaging was evaluated in a subset of participants at selected centers.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: The ITT-MRI population consisted of all randomized participants who participated in the MRI cohort and had evaluable Baseline MRI data. A multiple imputation process was used.
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid Injection | Placebo
Number analyzed (Participants) | 113 | 111
percentage of participants | 46.3 | 5.3
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection vs Placebo; If both primary endpoints were statistically significant, testing continued to the 2 secondary endpoints using the Bonferroni-Holm method. The smaller of the 2 p-values for the treatment difference was tested at the 0.025 level. If significant, testing proceeded for the remaining secondary endpoint at the 0.05 level. If the smaller p-value was > 0.025, the null hypothesis for the associated variable would not be rejected, and testing of the second endpoint would not proceed; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH method stratified by pooled study center; Risk Ratio (RR) = 8.541, 95% CI 2-sided [3.620 to 20.148] — A risk ratio greater than 1 favors deoxycholic acid injection treatment, and between 0 and 1 favors placebo

4. Secondary Outcome: Change From Baseline in Patient-Reported Submental Fat Impact Scale (PR-SMFIS)
Description: The PR-SMFIS assesses the impact of submental fat on self-perception of 6 emotional and visual characteristics related to the appearance of submental fullness (unhappy, bothered, self-conscious, embarrassed, look older, and look overweight) as evaluated by the participant. Each item is rated on an 11-point numeric scale from 0 to 10. Scores for the 6 items were averaged to generate a PR-SMFIS total scale score ranging from 0 to 10 where 0 is a positive outcome and 10 is a negative outcome. A negative change from Baseline indicates improvement.
Time Frame: Baseline and 12 weeks after last treatment (up to 32 weeks after first treatment)
Population: Intent-to-treat population; missing values were imputed using a multiple imputation process.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deoxycholic Acid Injection | Placebo
Number analyzed (Participants) | 256 | 250
units on a scale | -3.56 (2.793) | -1.16 (2.064)
Statistical Analysis 1: Comparison: Deoxycholic Acid Injection vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) model included treatment and Baseline PR-SMFIS total scale score

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 24 weeks after the last dose (up to 44 weeks after first treatment).
Description: The safety population consisted of all participants who received at least 1 injection of study drug. One participant was randomized to placebo, received deoxycholic acid injection at Visit 4 (Week 8), and was included in the deoxycholic acid injection arm for safety analyses.
Arm/Group | Deoxycholic Acid Injection | Placebo
Serious Adverse Events (participants affected / at risk) | 6/257 | 12/248
Other Adverse Events (participants affected / at risk) | 246/257 | 196/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection (N=257) | Placebo (N=248)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess oral (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Meningism (Nervous system disorders) | 1 | 0
Urethral disorder (Renal and urinary disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid Injection (N=257) | Placebo (N=248)
Injection site haematoma (General disorders) | 180 | 167
Injection site pain (General disorders) | 168 | 58
Injection site oedema (General disorders) | 136 | 54
Injection site anaesthesia (General disorders) | 172 | 11
Injection site swelling (General disorders) | 96 | 39
Injection site erythema (General disorders) | 46 | 25
Injection site induration (General disorders) | 47 | 4
Injection site paraesthesia (General disorders) | 33 | 8
Injection site nodule (General disorders) | 32 | 2
Injection site pruritus (General disorders) | 22 | 9
Nasopharyngitis (Infections and infestations) | 23 | 26
Headache (Nervous system disorders) | 19 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Study Agreement requires that the investigator or institution obtain written consent from Kythera prior to presenting and/or publishing results of this study.